CLINICAL TRIAL: NCT02849925
Title: Randomized Controlled Clinical Trial on the Treatment of Caries Lesions Using Resin or Glass Ionomer Sealants in Permanent Teeth
Brief Title: Sealing Microcavitated Carious Lesions
Acronym: SealCaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Talca (Other)
Responsible Party: Principal Investigator, Rodrigo A. Giacaman, Associate Professor, University of Talca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCTICDAS3/2015
Record Dates: First submitted 2016-07-21; First posted 2016-07-29 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Dental Caries
Keywords: Pit and Fissure Sealants; Caries; Glass ionomer; Resin
MeSH Terms: conditions — Dental Caries; Van der Woude syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glass Ionomer Sealant (Experimental): Sealants to arrest microcavitated caries. 75 microcavitated ICDAS 3 lesions will be sealed by the use of Glass ionomer sealant, EQUIA (GC) in first permanent molars.
  Interventions: Drug: Sealants to arrest microcavitated caries.
- Resin Sealant (Active Comparator): Sealants to arrest microcavitated caries. 75 microcavitated ICDAS 3 lesions will be sealed by the use of resin sealant, Clinpro (3M-ESPE) in first permanent molars
  Interventions: Drug: Sealants to arrest microcavitated caries.

INTERVENTIONS:
Drug: Sealants to arrest microcavitated caries. — Carious lesions will be treated by minimally invasive dentistry by the use of sealants instead of eliminating carious tissues and using conventional restorative materials.
  Other Names: Carious lesion arrest

SUMMARY:
This study aimed to test whether sealing microcavitated ICDAS 3 carious lesions in permanent molars may be arrested by sealing using two different types of materials; a glass ionomer and a resin sealant. A Randomized controlled clinical trial was designed. Children between 6 and 12 years old were recruited and a total of 150 ICDAS 3 lesions in first permanent molars were allocated to one of the two arms of the study. Clinical and radiographic lesion progression were the main outcome. Integrity of the material and retention were secondary outcomes. A follow up period of 24 months with check-ups at 6 and 12 months was considered.

DETAILED DESCRIPTION:
Background and problem statement. Traditionally, caries treatment has been based on restorative procedures performed by dentist using dental biomaterials. Besides its high cost, this canonical approach for caries therapy has very limited coverage and only a small proportion of the population can satisfy the high demand. The latter is especially critical in developing countries. Available evidence has shown that some caries lesions, either cavitated or non-cavitated, may be treated by the placement of sealants. This minimally invasive treatment is more cost-effective than the restorative approach and it allows better coverage. Sealants placed on the active lesions hamper lesion progression, most likely by inhibiting nutrient uptake of the invading associated microbiota. The most commonly used material in clinical practice is resin sealant. Despite its advantages and simplicity of use, this material is highly sensitive to contamination by saliva or other ubiquitous oral fluids. Furthermore, adhesion to enamel is compromised when this tissue is immature. This pitfall of the technique is particularly crucial when it comes to treating lesions in erupting molars in children. Hence, glass ionomer cement (GI) sealants emerge as a potential alternative to resin sealants. GI sealants are more suitable to be used under non-ideal clinical conditions, such as in the presence of humidity or on lesions of immature erupting molars. Although there exists vast evidence on the use of sealants as preventive agents, studies dealing with this biomaterial as a therapeutic agent for caries lesions are more limited and scarce. In regard to the material, only few clinical studies with unclear conclusions are available. This proposal, therefore, will seek to compare progression of caries lesions treated with either resin or GI sealants, in occlusal cavitated lesions (Code 3, ICDAS) of permanent molars of 6 to 12 year-old children.

Methodology. A randomized controlled clinical trial (RCT) is proposed. Once approved by the Bioethics Committee and after obtaining a signed informed consent from their parents, volunteer children will be invited to participate. Two hundred caries lesions (Code 3, ICDAS) will be randomized to one of the two arms of the study, resin or GI sealants. The materials chosen to conduct the study would be Concise and Ketac Molar, respectively, both from 3M, St. Paul, MN. Sample size was estimated using a 95% significance level. Based on the caries prevalence of the population and studies performed by the investigators, the number of volunteers was estimated to be about one hundred volunteers to gather the required two hundred lesions. Three evaluations will be conducted every six months until completion of eighteen month of follow-up. All the exams and controls will be performed at the Dental Clinics of the University of Talca by one trained and calibrated examiner. Sealants will be placed following manufacturer's instructions. Participants will be randomly allocated to either study arm, regardless of the clinical indication, so selection bias will be avoided. Material retention and lesion progression will be the primary end-point at each control. Likewise, caries incidence in untreated teeth will be a secondary outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* To have at least one ICDAS 3 lesion in first permanent molars
* To be systemically healthy

Exclusion Criteria:

* Not fully erupted first molars
* Structural defects in first molars, i.e., hypoplasia, fluorosis, MIH.
* Periodontal disease
* Orthodontic appliances
* Medication use

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of lesions that evidence progression by a higher ICDAS code. The score will be expressed as percentage of progression among all the treated lesions. | 24 months
  ICDAS 3 lesions will be followed and monitored for clinical and radiographic progression

SECONDARY OUTCOMES:
Percentage of sealants that were intact from the first intervention over time. | 24 months
  Sealants used will be monitored for integrity and retention
Percentage of sealants that were fractured or lost during the follow-up. | 24 months
  Sealants used will be monitored for integrity and retention

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Talca, No State, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz-Sandoval C, Gambetta-Tessini K, Giacaman RA. Microcavitated (ICDAS 3) carious lesion arrest with resin or glass ionomer sealants in first permanent molars: A randomized controlled trial. J Dent. 2019 Sep;88:103163. doi: 10.1016/j.jdent.2019.07.001. Epub 2019 Jul 2. PMID 31276747